CLINICAL TRIAL: NCT02320357
Title: Pilot Study Related to the Effect of Clopidogrel on Plasmatic Soluble CD40 Ligand During Systemic Lupus Erythematous
Acronym: CLOPUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2013/27
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Systemic Lupus Erythematous
Keywords: Platelet activation; CD40 ligand; CD154; Interferon alpha; clopidogrel
MeSH Terms: conditions — Hyper-IgM Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clopidogrel (Experimental)
  Interventions: Drug: Treatment by clopidogrel

INTERVENTIONS:
Drug: Treatment by clopidogrel — Peripheral blood will be obtained during the study

SUMMARY:
CD40 Ligand (CD40L) has been identified as a key feature in systemic lupus erythematosus (SLE) pathogenesis, a systemic autoimmune disease characterized by a multiorgan involvement. As platelets are a major source of soluble CD40L (sCD40L), we propose to study the effect of clopidogrel, a platelet inhibitor, on plasmatic sCD40L levels in SLE patients.

DETAILED DESCRIPTION:
Type I interferon (IFN) and CD40L have been identified as important in SLE pathogenesis (1). CD40L is now considered as a biomarker of lupus activity (4). Because platelets represent a major reservoir of CD40L, we previously studied the role of platelet derived CD40L in SLE pathogenesis (5). We showed that platelets from SLE patients were activated in vivo by circulating immune complexes composed of autoantibodies bound to self antigens through a Fc-gamma Receptor IIa (CD32)-dependent mechanism. Further, platelet activation correlated with severity of the disease and activated platelets formed aggregates with antigen-presenting cells including monocytes and plasmacytoid dendritic cells. In addition, activated platelets enhanced IFN-α secretion by immune complexes-stimulated plasmacytoid dendritic cells in vitro through a CD154-CD40 interaction. In lupus prone mice, depletion of platelets or administration of the clopidogrel improved all measures of disease activity and overall survival. In this pilot study the treatment of the research is clopidogrel given at the dose of 75mg once a day. For the features of the treatment, its contraindications, its disruption in case of side effects cf to annex 1. Clopidogrel associated with the usual treatment of patients will be given for 12 weeks, the follow up of patients will be 16 weeks, all side effects occurring during this period will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE according to revised criteria of American College of Rheumatology
* Being affiliated to health insurance
* Having signed an informed consent (later than the day of inclusion and before any examination required by research)

Exclusion Criteria:

* > 20mg/day of prednisone equivalent for > 7 days 30 days before the pre-inclusion.
* Diseases flare 3 months before the inclusion. A disease flare is defined by an increase of SLEDAI score >3 and or a change of the immunosuppressive treatment and or an increase of steroids dose.
* Is treated or has received 3 months before the pre-inclusion steroids pulses or intravenous immunoglobulins.
* Renal involvement that could required a kidney biopsy.
* Required surgery in the next 12 weeks.
* Has been treated by cyclophosphamide 3 months before the pre-inclusion.
* Has been treated by biotherapy 6 months before the pre-inclusion.
* Contraindication to clopidogrel (annex 1).
* History of cancer except healed basal cell carcinoma.
* History of severe hemorrhage
* Disease exposing to hemorrhage
* Associated antiphospholipid syndrome
* Pregnant or breastfeeding women
* No contraception for women of childbearing age
* Severe hypertension
* Ongoing statin, non-steroidal anti-inflammatory, antiplatelet and anticoagulant drugs.
* Being under guardianship
* Patient participating at an other biomedical research with an exclusion period at the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Measurements of plasmatic sCD40L levels | 12 weeks afther the inclusion (D0)

SECONDARY OUTCOMES:
Measurements of plasmatic sCD40L levels | At 1 month before the inclusion (M-1) and at 24 hours, 7 days, 4, 8 and 16 weeks after the inclusion (D0)
Measurements of IFN inducible genes by RT-PCR in circulating monocytes | At the inclusion (D0) and 12 weeks after the inclusion (D0)
Measurements of platelet activation markers by flow cytometry | 12 weeks afther the inclusion (D0)
Measurements of platelet/circulating mononuclear cells aggregates by flow cytometry | At 7 days and 12 weeks after the inclusion (D0)
Measurements of T lymphocytes activation by flow cytometry | At 7 days and 12 weeks after the inclusion (D0)
Rate of haemorrhagic side effects during the follow up | At 24 hours, 7 days, 4, 8, 12 and 16 weeks after the inclusion (D0)
Measurements of inflammation markers, antiantibodies levels, complement fractions | At 24 hours, 7 days, 4, 8, 12 and 16 weeks after the inclusion (D0)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DUFFAU, MD, Principal Investigator — University Hospital Bordeaux, France; Rodolphe THIEBAUT, Prof, Study Chair — University Hospital Bordeaux, France
Locations (3):
- France (3):
  - Service de Médecine Interne et maladies Infectieuses - Hôpital Saint-André, Bordeaux
  - Service de Médecine Interne, Limoges
  - Service de Médecine Interne et Immunopathologie, Toulouse